CLINICAL TRIAL: NCT04253171
Title: Balloon Lithoplasty for Preparation of Severely Calcified Coronary Lesions Before Stent Implantation - a Nationwide Randomized Trial (BALI)
Brief Title: Balloon Lithoplasty for Preparation of Severely Calcified Coronary Lesions
Acronym: BALI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Abbott (Industry); Shockwave Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Niels Thue Olsen, Primary Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19051822
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Percutaneous Coronary Intervention; Coronary Artery Calcification; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Lithotripsy

STUDY DESIGN:
Intervention Model Description: Investigator-initiated 1:1 randomized, controlled, multinational, superiority trial.
Who Masked: Outcomes Assessor
Masking Description: The primary outcome will be assessed by a blinded clinical events adjudication committee and by a blinded OCT core laboratory analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lithoplasty lesion preparation (Active Comparator): Balloon lithoplasty will be used as lesion preparation.
  Interventions: Device: Lithoplasty
- Conventional lesion preparation (Active Comparator): Conventional and modified balloons will be used as lesion preparation.
  Interventions: Device: Conventional

INTERVENTIONS:
Device: Lithoplasty — The lithoplasty balloon should be utilized as early as possible. If it is necessary for passage of the lithoplasty balloon, the lesion may first be predilated with an undersized conventional balloon, non-compliant or semi-compliant. If passage of the lithoplasty balloon is still not possible, it is recommended to perform rotational atherectomy with a small burr size.
  The lithoplasty balloon is sized 1:1 to reference diameter. Lithoplasty is performed with the balloon dilated at 4 atmospheres, and 10 shocks are delivered, after which the balloon is expanded to 6 atmospheres for 30 seconds, and then deflated. Up to 8 series of balloon expansion/deflation can be delivered in this manner if necessary, and several balloons may be used for long lesions.
  Other Names: Shockwave; Lithotripsy
  Arms: Lithoplasty lesion preparation
Device: Conventional — Lesion preparation is performed starting with conventional balloons, non-compliant or semi-compliant. Unless fully satisfactory dilatation is achieved with conventional balloons, it is recommended to also use modified balloons (scoring balloons, cutting balloons). If balloons cannot be passed or if dilatation is inadequate, the lesion may first be predilated with an undersized conventional, non-compliant, or semi-compliant balloon. If necessary, rotational atherectomy with a small burr size can be used to facilitate adequate balloon preparation.
  Arms: Conventional lesion preparation

SUMMARY:
Severely calcified coronary stenoses are difficult to treat with percutaneous coronary intervention (PCI) using current techniques and there is little specific evidence on how to best treat these cases. It is hypothesized that balloon lithoplasty is superior to conventional balloons for lesion preparation of severely calcified coronary lesions before stent implantation in terms of procedural failure and 1-year target vessel failure.

DETAILED DESCRIPTION:
Severely calcified coronary stenoses are difficult to treat with percutaneous coronary intervention (PCI) using current techniques. Severe calcifications make it difficult to sufficiently prepare lesions before stenting, to advance stents, and to achieve full stent expansion. There is increased risk of vessel dissection and perforation with angioplasty on severely calcified lesions, and long-term outcomes of PCI are adversely affected. Because severely calcified lesions are often excluded from interventional studies, there is little specific evidence on how to best treat these cases. Only a few randomized studies have specifically explored this question, focusing on the use of rotational atherectomy

Recently, the technique of balloon-based lithoplasty was made commercially available. With this technique, calcifications are cracked with the creation of high-frequency pressure oscillations in a special angioplasty balloon. Standard techniques are used to deliver and dilate the balloon. The method was developed for treatment of otherwise non-dilatable lesions, and first reported results have been encouraging. The lithoplasty device used in the current study (Shockwave IVL, Shockwave Medical, CA, USA) has received CE-mark and post-approval safety has recently been confirmed for treatment of severely calcified coronary lesions in patients.

Besides obvious benefits in non-dilatable lesions for which interventional cardiologists have few other options, it is possible this technique could change the way all severely calcified lesions are treated. Balloon lithoplasty could theoretically crack plates of calcium in the vessel wall in an orderly fashion, which could lead to safer and quicker preparation of severely calcified lesions. Furthermore, a better softening of vessel wall calcium could allow full and symmetric expansion of coronary stents, which could lead to better long-term stent patency.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 90 years
* Stable coronary heart disease or non-ST elevation acute coronary syndrome
* PCI planned in severely calcified, non-occluded, de-novo lesion in native vessel. Definition of severe calcifications (minimum 1 of 3 (i-iii)); i. Angiography: Radioopacities of the vessel wall visible on cine images before contrast injection on both sides of the vessel lumen in more than one projection. ii. OCT (before lesion preparation): Maximum calcium 1) angle >180 degrees AND 2) thickness 0.5mm, AND 3) longitudinal length >5m m. iii. IVUS (before lesion preparation): Maximum calcium angle >270 degrees.
* Functional evidence of ischemia (non-invasive stress test or fractional flow reserve) in the target vessel territory or stenosis ≥ 90% by visual estimate
* Target vessel reference diameter visually estimated at 2.5-4 mm with ability to pass a 0.014" guidewire across lesion
* Ability to tolerate dual antiplatelet therapy
* Informed consent

Angiographic exclusion criteria:

* Unprotected left main stenosis
* Chronic total occlusion
* Severely calcified bifurcated lesion with expected need to use two stent technique
* Coronary artery dissection

Clinical exclusion criteria

* ST-segment elevation acute myocardial infarction
* Planned later revascularization in non-study lesions
* Planned cardiovascular intervention within 30 days after study intervention
* Clinical instability including decompensated heart disease
* Life expectancy of less than 1 year
* Active peptid ulcer or upper gastrointestinal bleeding within 6 months
* Ongoing systemic infection

Paraclinical exclusion criteria

* Left ventricular ejection fraction <35 %
* Renal function with eGFR <30 mL/min
* Pregnant or nursing

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with combined outcome of strategy failure | 1 year
  Failed stent delivery, residual area stenosis ≥ 20% (OCT-assessed) after PCI, or target vessel failure.
  Residual area stenosis will be defined as [1 - in-stent minimal lumen area/reference area]. The reference area will be calculated by averaging the proximal and distal reference areas, which will be determined by measuring the lumen contours on most healthy-looking frame of the final OCT in the 0-5 mm edge segments. If a reference cannot be measured on the final OCT, it will be measured on a pre-stent OCT or by using quantitative coronary angiography if pre-stent OCT is unavailable. Target vessel failure will be defined as cardiac death, target vessel-related myocardial infarction, or clinically driven target vessel revascularization). Failed or no stent delivery is defined as failure to deliver and deploy 1 or more coronary stents to cover the intended length of the intended target lesion.

SECONDARY OUTCOMES:
Number of patients with composite and components of in-hospital major adverse cardiac events (MACE) | In-hospital
  Cardiac death, Any myocardial infarction, Stroke
Number of patients with composite and components of major adverse cardiac events (MACE) | 1 year
  Cardiac death, Any myocardial infarction, Stroke
Number of patients with in-hospital procedure-related adverse events | In-hospital
  Periprocedural myocardial infarction, Coronary dissection (beyond intended by lesion preparation), Coronary perforation/rupture
Number of patients with components of the primary outcome | 1 year
  Failed stent delivery, Residual area stenosis >20% (OCT-assessed) after PCI, Target vessel failure
Number of patients with components of target vessel failure | 1 year
  Cardiac death, Target vessel-related myocardial infarction, Clinically driven target vessel revascularization
OCT outcomes at index procedure | During procedure
  Stent expansion
OCT outcomes at 1 year procedure | 1 year
  In-stent late lumen loss

CONTACTS AND LOCATIONS:
Overall Officials: Niels Thue Olsen, MD, PhD, Principal Investigator — Herlev and Gentofte Hospital
Locations (9):
- University Hospital Leuven, Leuven, Belgium
- Denmark (6):
  - Gentofte University Hospital, Gentofte Municipality, Copenhagen
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital Skejby, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde Sygehus, Roskilde
- North-Estonia Medical Center, Tallinn, Estonia
- Trondheim University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kristensen AT, Christiansen EH, Holm NR, Kelbaek H, Engstrom T, Veien K, Raungaard B, Kleveland O, Bennett J, Laanmets P, Jakobsen L, Havndrup O, Lonborg JT, Ahlehoff O, Iversen A, Vatwani AK, Stottrup NB, Jensen LO, Christensen MK, Haahr-Pedersen SA, Charlot MG, Gabriel EE, Olsen NT. Balloon Lithotripsy Added to Conventional Preparation Before Stent Implantation in Severely Calcified Coronary Lesions. JACC Cardiovasc Interv. 2025 Nov 18:S1936-8798(25)02480-X. doi: 10.1016/j.jcin.2025.09.028. Online ahead of print. PMID 41400597

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04253171/SAP_001.pdf